CLINICAL TRIAL: NCT03244553
Title: Treatment of Dysphagia and Ineffective Esophageal Motility With Prucalopride: A Pilot Study
Acronym: IEMPru
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Michelle Buresi, Principal Investigator, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGMC-Pru-02
Record Dates: First submitted 2017-08-01; First posted 2017-08-09 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Ineffective Esophageal Motility; Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — prucalopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active intervention (Experimental): Prucalopride for 5 days. Dosage: day 1 2mg, days 3-5 4mg
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: Prucalopride — 5 day treatment

SUMMARY:
This study will test prucalopride (a prokinetic drug currently approved by Health Canada for treatment of constipation) as a treatment for Ineffective Esophageal Motility (IEM). Adult patients with previously diagnosed IEM will be invited to participate by the investigators. The participants will take the study medication for 5 days and on the final day of medication undergo an esophageal manometry procedure at the Calgary Gut Motility Centre to measure esophageal function. Symptoms and side effects will be tracked at baseline and on Day 5.

DETAILED DESCRIPTION:
As part of the standard clinical evaluation of our department, all patients presenting to the Calgary Gut Motility Centre with dysphagia routinely undergo a thorough clinical assessment including history taking and physical examination. Depending on their presentation, further evaluation may include upper endoscopy, barium swallow, esophageal manometry, and pH testing.

Patients meeting inclusion and exclusion criteria will receive prucalopride for 5 days total, with 2mg on day 1, then 4mg on days 2 to 5. On day 5 of the intervention, patients will undergo esophageal manometry. Patients will also complete a symptoms questionnaire for assessment of dysphagia symptoms and the EQ-5D questionnaire for assessment of global quality of life at baseline and on day 5 of prucalopride treatment.

Full research ethics approval will be obtained prior to commencement of the study. Participants will be recruited from patients completing esophageal manometry at the South Health Campus. Patients who have provided consent to be contacted for research studies and who have dysphagia and findings of ineffective esophageal motility (IEM) on manometry will be contacted by the study investigators. The results of their esophageal manometry will be reviewed with them, and the study will be described to them. If the patient is interested in study participation, then study investigators will arrange for the patient to come to the South Health Campus to review the study in detail prior to obtaining informed consent. Thirty patients will be enrolled in this study.

Patients who meet all inclusion and exclusion criteria will be enrolled. Once enrolled, the participants will be asked to complete a symptom and quality of life questionnaire. They will receive the prucalopride pills, to be taken for 5 days with the following instructions: Day 1, take 1 tablet (2 mg), on days 2 through 4, take 2 tablets (4mg) and on day 5, take 2 tablets 1 hour prior to the second scheduled study appointment. On day 5, the patient will be scheduled at South Health Campus for esophageal manometry. Patients will also be asked to complete a post-treatment symptom and quality of life questionnaire at that time.

ELIGIBILITY:
Inclusion Criteria:

* Symptom of dysphagia
* Esophageal findings consistent with ineffective esophageal motility (IEM), defined as per the Chicago Classification as ≥50% ineffective swallows. Ineffective swallows include both failed swallows, defined by an average distal contractile integral (DCI) <100mmHg*cm*sec, and weak swallows, defined by an average DCI >100 but <450mmHg*cm*sec
* Normal endoscopy
* If female of childbearing potential, a negative urine pregnancy test administered 1 day prior to taking the study medication (prucalopride)
* Able to provide informed consent

Exclusion Criteria:

* Clinical evidence (on history, physical exam, or investigations) of significant cardiovascular, respiratory, gastrointestinal, hepatic, hematological, renal, neurological, or psychiatric comorbidities that may interfere with the objectives of the study and/or pose safety concerns, including pregnancy and breastfeeding
* History of cardiovascular disorder including myocardial infarction, life-threatening arrhythmias, pacemaker or defibrillator
* Estimated GFR <30, documented within 6 months preceding study entry
* Blood electrolytes (Na, K, CL) measured within past 6 months outside of normal reference ranges
* Uncontrolled gastroesophageal reflux disease on pH testing (DeMeester score >14.7)
* Established esophageal motility disorder, including but not limited to achalasia, spastic disorders, Esophagogastric junction (EGJ) outflow obstruction, and absent contractility
* History of gastrointestinal surgery, including hiatal hernia repair and/or fundoplication, or any major surgery in the 3 months preceding study entry
* Use of narcotics or prokinetic treatments that cannot be stopped prior to study entry
* Use of laxatives that cannot be stopped prior to study entry
* Use of tricyclic antidepressants at a dose of >25 mg daily (stable doses of SSRIs/ SNRIs are permitted)
* Use of macrolide antibiotics (non-macrolide antibiotics are permitted)
* Participation in clinical trial with prokinetic treatment in the 30 days preceding study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Change in number of successful swallows | Baseline and on day 5 of treatment
  Esophageal Manometry

SECONDARY OUTCOMES:
Change in Dysphagia Questionnaire Score | Baseline and on day 5 of treatment
  Mayo 30
Change in EQ-5D Score | Baseline and on day 5 of treatment
  Quality of life/health related

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Buresi, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No